CLINICAL TRIAL: NCT01608217
Title: Efficacy and Safety of Delta-9-tetrahydrocannabinol (∆9-THC) in Behavioural Disturbances and Pain in Dementia
Brief Title: Delta-THC in Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Health Valley, Netherlands (Network)
Responsible Party: Principal Investigator, Marcel Olde Rikkert, Prof. dr. Marcel Olde Rikkert, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GER001-02-02; 2011-005289-39 (EudraCT Number); NL38617.091.12 (Registry Identifier: toetsingonline.com)
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Behavioural Disturbances; Pain; Dementia; Alzheimer's Dementia; Vascular Dementia
Keywords: Behavioural disturbances; Pain; Dementia; Alzheimer's dementia; Vascular dementia; THC; Cannabis
MeSH Terms: conditions — Mental Disorders; Pain; Dementia; Alzheimer Disease; Dementia, Vascular; Marijuana Abuse | interventions — Dronabinol; nabiximols; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Namisol (Active Comparator): Namisol is a tablet containing delta-9-tetrahydrocannabinol, the main cannabinoid from Cannabis sativa L. Namisol is added to a standardized treatment with acetaminophen.
  Interventions: Drug: delta-9-tetrahydrocannabinol (delta-THC); Drug: Acetaminophen
- Placebo (Placebo Comparator): The control product is placebo, consisting of a tablet with similar appearance and taste of the test product. Placebo is added to a standardized treatment with acetaminophen.
  Interventions: Drug: Placebo; Drug: Acetaminophen

INTERVENTIONS:
Drug: delta-9-tetrahydrocannabinol (delta-THC) — delta-THC 1.5 mg (tablet)three times daily for a period of 3 weeks.
  Other Names: Namisol; Cannabis; ECP002A
  Arms: Namisol
Drug: Placebo — placebo (tablet) three times daily for a period of three weeks.
  Arms: Placebo
Drug: Acetaminophen — Acetaminophen 1000 mg three times daily for a period of 3 weeks
  Other Names: Paracetamol
  Arms: Namisol
Drug: Acetaminophen — Acetaminophen 1000 mg three times daily for a period of three weeks
  Other Names: Paracetamol
  Arms: Placebo

SUMMARY:
This is a phase II, randomized, placebo-controlled, double-blind, parallel-group, multicentre study to the efficacy and safety of low dose delta-9-THC in behavioural disturbances and pain in patients with mild to severe dementia, when added to an analgesic treatment with acetaminophen.

It is hypothesized that Namisol® will lead to more behavioural disturbances than placebo, when added to an analgesic treatment with acetaminophen, and as measured by a change in Neuropsychiatric Inventory (NPI) score, after a three week treatment period.

It is expected that this will be due, primarily, to psychoactive effects of Namisol® and secondary to a reduction in pain sensation (as measured with VRS and PACSLAC-D). It is expected that a reduction in NPS will positively affect quality of life and lead to better functioning in daily living.

DETAILED DESCRIPTION:
There is a high prevalence of behavioural disturbances (NPS) in persons with dementia. Persistent pain complaints can be a cause of NPS. Unfortunately, there is a lack of appropriate drugs for treating both these problems. This and positive suggestions from preliminary clinical studies with THC on NPS and directly fuel the study presented here.

This will be a phase II study in which the efficacy and safety of Namisol® (a tablet with THC) on behavioural disturbances, such as agitation, aggression and motor disturbances in dementia patients will be evaluated.

Secondary study objectives are :

2. To evaluate the efficacy of Namisol® on other secondary outcome measures, such as quality of life and functioning in daily activities.

3. To evaluate safety of Namisol® as assessed with physical examination, effects on cognitive functioning and adverse event monitoring.

4. For the subgroup of subjects suffering from pain: to evaluate the efficacy of Namisol® pain intensity

It is hypothesized that Namisol® will lead to more reduction in behavioural disturbances than placebo, when added to an analgesic treatment with acetaminophen, and as measured by a change in Neuropsychiatric Inventory (NPI) score, after a three week treatment period. It is expected that this will be due, primarily, to psychoactive effects of Namisol® and secondary to a reduction in pain sensation (as measured with VRS and PACSLAC-D). It is expected that a reduction in NPS will positively affect quality of life and lead to better functioning in daily living

This is a randomized placebo-controlled double-blind parallel-group multicentre study.

Subjects who appear to fulfill the eligibility criteria are informed about the study. After signing informed consent by the subject and/or caregiver, a screening visit will take place. Subjects who are eligible for participation enter a wash-out period, for discontinuation of their own analgesic medication (if applicable). Subjects will be randomly allocated to receive one of the two interventions (Namisol® 1.5 mg + acetaminophen 1000 mg three times daily, or placebo + acetaminophen 1000 mg three times daily) for a double-blind intervention period of three weeks. After two weeks the primary outcome measure (NPI) is assessed by a telephone interview with the caregiver. Subjects visit the site twice (at baseline and after three weeks treatment) for assessments of the outcome parameters, including the NPI. For the purpose of compliance and safety, there will be a weekly phone call, performed by the researcher. After completion of this period subject's own analgesic treatment will be restarted (if applicable). After a follow up phase of two weeks, the subject is contacted by telephone for assessment of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject has possible or probable dementia, type Alzheimer, vascular or mixed type dementia, according to the criteria of NINCDS-ADRDA/NINCDS-AIREN or based on an expert panel decision.
* Clinical Dementia Rating (CDR) score 1 to 3 (mild to severe dementia).
* Age ≥ 40 years.
* Clinically relevant behavioral disturbances existing at least one month prior to screening, defined as a score of ≥ 10 on the NPI, including presence of the domain agitation/aggression or motor disturbance.
* Women should be in the postmenopausal phase.
* Availability of an informal or formal caregiver, being in touch with the subject at least twice a week.
* Informed consent by the subject and subject's informal caregiver.
* If applicable: subject is willing to stop his/her own pain medication, for the duration of the study.

Exclusion criteria:

* Dementia other than AD, VaD or AD/VaD
* Major psychiatric disorder such as: major depression according to DSM IV within 6 months prior to randomization, history of psychosis or mania, current hallucinations and/or delirium, current suicidal ideation or major anxiety disorder.
* History of, or current drug abuse.
* Current alcohol abuse or unwillingness to use no more than 2 alcoholic consumptions daily or raised gamma-glutamine transpeptidase and alkaline phosphatase .
* Clinical or biochemical evidence of liver disease (ALT or AST ≥ twice the upper limit of normal) or known allergy to acetaminophen.
* Severe (and/or unstable) concomitant or intercurrent illness, such as seizure, arrhythmias requiring other drugs than a beta blocker or digoxin (except sinus arrhythmia and atrial fibrillation), unstable angina pectoris, heart failure NYHA III or IV, and severe concomitant illness that requires treatment changes.
* Known or suspected sensitivity to cannabinoids.
* Lactosis intolerance.
* Frequent falling due to orthostatic hypotension.
* Use of tricyclic antidepressants (TCA), fluoxetine and/or carbamazepine.
* Changes in dosage of antipsychotics, benzodiazepines or cholinesterase inhibitors within 2 weeks prior to intervention.
* Participation in any other study other than the descriptive 'Parelsnoer' study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (NPI) | Screening, baseline, T= 2 weeks (by telephone interview) and T=3 weeks
  The NPI has been accepted as the standard measure of NPS in most clinical trials, due to high validity, good inter-rater reliability, high internal consistency and its sensitivity to drug treatment effects. In clinical practice as well as clinical research the NPI is the most commonly used instrument to assess behavioral changes. The NPI evaluates 12 behavioral domains. The frequency and severity of these behaviors is scored by the informal caregiver.

SECONDARY OUTCOMES:
Pain Assessment Checklist for Seniors with Limited Ability to Communicate Dutch version (PACSLAC-D) | baseline (T = 0) and T= 3 weeks
  The PACSLAC-D is a brief version of Pain Assessment Checklist for Seniors with Limited Ability to Communicate in Dutch to observe pain related behavior It consists of 24 items, separated in three subscales (facial and vocal expressions, resistance/defense, social-economical aspects/mood). This scale is one of the few instruments in which the items are specifically geared towards elderly with dementia.
Caregiver Clinical Global Impression of Change (CCGIC) | baseline (T=0), T= 2 wks (by telephone interview) and T=3 wks
  The CCGIC is a 7-point Likert scale that assesses global change from baseline. The scale ranges from 1 ('very much improved') to 7 ('very much worse'). It has been frequently used in several psychopharmacological trials and in early clinical trials for antidementia drugs. When the caregiver rates the subject as changed compared to baseline, this change is, by definition, clinically meaningful.
Cohen-Mansfield Agitation Inventory (CMAI) | baseline (T=0) and T= 3 weeks
  The CMAI is selected to assess agitation and aggression. It is an internationally validated instrument, specifically developed to measure behavioral disturbance in people with dementia
Quality of Life-Alzheimer's Disease Scale (QoL-AD) | baseline (T=0) and T= 3 weeks
  The QoL-AD is a 13 -item self-report scale, using four-point Likert-scales, but can also be completed in conjunction with the interviewer. It is developed for assessment of quality of life in subjects with mild to moderate severe dementia, but there is also evidence for reliability in severe dementia.
Barthel Index | baseline (T=0) and T = 3 weeks
  The Barthel Index was originally developed to assess disability in patients with neuromuscular and musculoskeletal conditions receiving rehabilitation, but is also recommended for functional assessment in elderly. Barthel Index is an easy to conduct, 10-item scale which scores several primary activities of daily living.
Paired Associates Learning test Wechsler Memory Scale Revised(PAL WMS-R) | baseline (T = 0) and T = 3 weeks
  The PAL is a WMS subtest for assessment of episodic memory function. The PAL is sensitive to midtemporal lobe dysfunction and therefore suitable for assessment of effects of THC on hippocampal functioning. This test entails the presentation of 10 pairs of common words that have to be remembered (6 semantically related and 4 unrelated pairs). After presentation of the word pairs, the researcher reads aloud the first word of each pair, which has to be completed by the subject, thereby assessing the capacity to recall.
Safety assessments | screening, baseline (T=0), T= 3 weeks. AE and compliance during telephone calls at T= 1week, T= 2 weeks and T= 5 weeks (follow up phone call)
  Safety will be assessed by physical examination, including vital signs and internal examination. On indication extended physical (internal and neurological) examination or diagnostic tests can be performed. An ECG will be performed in all subjects during every visit. The occurrence of (serious) adverse events will be monitored, from first administration of study medication onwards. Weekly telephone calls are scheduled using a THC-specific symptom checklist to assess possible adverse events
Verbal Rating Scale (VRS) | screening, baseline, T= 3 weeks, follow up (T= 5 weeks) and daily in a medication diary
  The VRS is an ordinal self-reporting scale for assessment of pain intensity. It is a 6-point scale consisting of a list of phrases that describe increasing levels of pain intensity. The subject selects that phrase best characterizing his/her pain intensity at that moment. In agreement with the Interdisciplinary Consensus Statement on Assessment of Pain in Older Persons the VRS is chosen as the self-reporting assessment method for pain intensity in this group with mild to moderate impaired cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Olde Rikkert, prof. dr., Principal Investigator — Radboud University Medical Center Nijmegen; Willem Verhoeven, Prof. dr., Principal Investigator — Vincent van Gogh voor Geestelijke Gezondheidszorg
Locations (2):
- Netherlands (2):
  - Radboud university medical center, department of Geriatrics, Nijmegen, Gelderland
  - Vincent van Gogh Institute for Psychiatry, department of Elderly, Venlo, Limburg

REFERENCES:
- [Derived] Bosnjak Kuharic D, Markovic D, Brkovic T, Jeric Kegalj M, Rubic Z, Vuica Vukasovic A, Jeroncic A, Puljak L. Cannabinoids for the treatment of dementia. Cochrane Database Syst Rev. 2021 Sep 17;9(9):CD012820. doi: 10.1002/14651858.CD012820.pub2. PMID 34532852
- See also: Dementia — http://www.nlm.nih.gov/medlineplus/dementia.html
- See also: Tetrahydrocannabinol — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0001972083&QV1=TETRAHYDROCANNABINOL
- See also: Cannabis — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0008063147&QV1=CANNABIS